CLINICAL TRIAL: NCT06300840
Title: Use of a Vibrotactile Feedback Belt in People With Chronic Disabling Unilateral Vestibular Hypofunction: a Single-case Experiment
Brief Title: Vibrotactile Feedback Belt in Patients With Unilateral Vestibular Hypofunction (UVH)
Acronym: VIBE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanna van Eijsden (Other)
Responsible Party: Sponsor-Investigator, Hanna van Eijsden, clinical investigator, Gelre Hospitals
Organization: Gelre Hospitals (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2023_49; NL84562.075.23 (Other: METC ISALA)
Record Dates: First submitted 2024-02-13; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Vestibular Disorder
Keywords: vibrotactile feedback
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Intervention Model Description: Single-case-experiment (SCE) with a reversal design and with randomization of phases.
Who Masked: Outcomes Assessor
Masking Description: Data-analyst and test-observer are masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline (No Intervention): Wearing no Balancebelt.
- Sham condition (Sham Comparator): Wearing the BalanceBelt while it is switched off
  Interventions: Device: BalanceBelt
- Intervention (Experimental): Wearing the BalanceBelt while it is switched on
  Interventions: Device: BalanceBelt

INTERVENTIONS:
Device: BalanceBelt — The vibrotactile belt (i.e., Elitac BalanceBelt®) supports patients with severe balance disorders by substituting the missing balance information with vibrations (haptic feedback).
  Arms: Intervention; Sham condition

SUMMARY:
The goal of this clinical trial is to study the impact of a continuous vibrotactile feedback belt on balance, (fear of) falling, fatigue and overall functioning in participants with chronic disabling unilateral vestibular hypofunction.

The main questions it aims to answer are: • does wearing a vibrotactile feedback belt during waking hours for a week improve sense of balance and mobility, fear of falling, fatigue and overall functioning • does wearing a vibrotactile feedback belt influence static and dynamic balance and gait performance during balance and gait testing.

Participants will goes through different phases in an randomized order; a baseline phase, a sham phase (i.e., wearing the BalanceBelt while it is switched off) and an intervention phase (i.e., wearing the BalanceBelt while it is switched on).

It is expected that, just as with patients with bilateral loss of the balance organ, patients with a unilateral loss will also benefit from the BalanceBelt.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with severe unilateral vestibular dysfunction (i.e., a gain below 0.6 of the affected side and a gain between 0.8 and 1.1 of the contralateral side measured by the video-Head Impulse Test (vHIIT)).
* Duration of dizziness complaints >3 months (i.e. chronic dizziness).
* Self-reported imbalance with a fear of falling and/or actual falls.
* Is able to walk (with or without a walking aid).
* Self-reported overall Mobility and Balance Score (MBS) of 3-5 points
* Motivated to try the BalanceBelt.
* Provides written informed consent.

Exclusion Criteria:

* Age < 18 years
* Presence of neurological, psychiatric or orthopaedic disorders, Persistent postural-perceptual dizziness (PPPD), reduced proprioceptive sensitivity or impaired vision which influences the postural stability.
* Not able to understand instructions and questionnaires in Dutch
* Not able/willing to visit Gelre Hospital Apeldoorn for necessary visits.
* Wheelchair bound at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Mobility and Balance Score (MBS) | Daily for 7 weeks
  The MBS is a rating given by the patient on a scale ranging from 0 to 10, as a subjective grading of his or her overall mobility and balance in daily life. Where a higher score means a better score.

SECONDARY OUTCOMES:
General functioning | Daily for 7 weeks
  Numeric rating scale (NRS), rang 0-10, where a higher score means a better outcome.
physical activity_NRS | Daily for 7 weeks
  Numeric rating scale, rang 0-10, where a higher score means a better outcome.
physical activity_steps | Daily for 7 weeks
  Number of steps a day
Fear of falling | Daily for 7 weeks
  Numeric rating scale, rang 0-10, where a higher score means a better outcome.
fatigue | Daily for 7 weeks
  Numeric rating scale, rang 0-10, where a higher score means a better outcome.
falls | Daily for 7 weeks
  number of actual falls and near falls
structured interview on compliance on wearing the Balancebelt(R) | Daily for 7 weeks
  compliance on wearing the Balancebelt(R)
Questionnaire: vestibular activity avoiding instrument (VAAI) | At baseline and at the end of the study (8 weeks)
  vestibular activity avoiding instrument, score range 0-54, higher score means worse outcome.
Questionnaire: Dizziness handicap inventory (DHI) | At baseline and at the end of the study (8 weeks)
  Dizziness handicap inventory, score range 0-100, higher score means worse outcome.
modified Clinical Test of Sensory Interaction on Balance (mCTSIB) | At baseline and at the end of the study (8 weeks)
  modified Clinical Test of Sensory Interaction on Balance
Dynamic Gait Index (DGI) | At the baseline and at the end of the study (8 weeks)
  Dynamic Gait Index, score 0-24, higher score means better outcome
Timed up and Go test (TUG) | At baseline and at the end of the study (8 weeks)
  Timed up and Go test

OTHER OUTCOMES:
age | Baseline
  in years
time since onset of the vestibular hypofunction | Baseline
  in months or years
cause of vestibular hypofunction | Baseline
  etiology
Structured interview on vestibular rehabilitation | Baseline
  previous experience with vestibular rehabilitation (types of intervention, number of therapie sessions, benefit)
outcome of the vestibular function tests | Baseline
  results of available video-Head Impulse Test (vHIT) or caloric testing
Structured interview on participating in the research | At the end of the study (8 weeks)
  experience of the research
Structured interview on the overall experience with the Balancebelt(R) | At the end of the study (8 weeks)
  evaluation of the Balancebelt(R)

CONTACTS AND LOCATIONS:
Overall Officials: Tjasse Bruintjes, PhD, Principal Investigator — Gelre Hop
Locations (1):
- Gelre Hospitals, Apeldoorn, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No